CLINICAL TRIAL: NCT06844890
Title: Depression Inventory for Maintenance Hemodialysis Patients: A Cross-Cultural Adaptation and Psychometric Evaluation in Turkey
Brief Title: Depression Inventory for Maintenance Hemodialysis Patients
Acronym: Depression
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul University
Other Study IDs: ATADEK-2022/06
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Depression; Hemodialysis Complication; Management; Risk Behavior
Keywords: depression; dialysis; management
MeSH Terms: conditions — Depression; Risk-Taking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression is frequently seen among hemodialysis patients; however, it causes an impaired quality of life, a decrease in adherence to treatment, and an increase in hospitalization and mortality rate. It has been stated in the literature that the prevalence rate of depression in hemodialysis patients varies between 25-73%. Despite its high prevalence rate and adverse effects, it has been revealed that only a low rate of patients with depressive symptoms are diagnosed and treated. This is primarily associated with the fact that depressive symptoms in patients are not adequately recognized and examined.

DETAILED DESCRIPTION:
Depression is assessed through structured clinical interviews or diagnostic scales. Structured clinical interviews are often regarded as the "gold standard" for the diagnosis of depressive disorders, since they are based on specific diagnostic criteria. However, since it is not always possible for patients to be evaluated by a psychiatrist, some scales are used instead. Even though these scales are not a diagnostic criterion, they are helpful in identifying patients at risk . However, screening may also result in false negatives, where cases of depression are not detected and, consequently, go untreated. Patients with kidney failure differ from the general population because they experience higher rates of comorbid depression. Indeed, there is a clear need for more effective screening tools for patients undergoing hemodialysis, given the wide variation in depression screening methods and the absence of a gold-standard assessment tool tailored to this specific population. Developing an easily administered, disease-specific self-report measure for depression could prove to be highly beneficial. There is only one study that has examined a depression tool specifically designed for patients on maintenance dialysis, known as the Depression Inventory-Maintenance Hemodialysis (DI-MHD)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients who were receiving hemodialysis treatment for at least three months
* Patients could communicate in Turkish
* Patients who agreed to participate in the study were included in the study.

Exclusion Criteria:

* Patients who suffered from psychiatric disorders such as chronic psychosis and were previously diagnosed with depression were excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taking hemodialysis therapy in dialysis unit
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Predict of depression risk with questionnare | Up to 15 days
  Depression Inventory for Maintenance Hemodialysis Patients The inventory, developed by the researchers consists of 17 items. In this four-point likert type scale; items are rated as never: 1 point, sometimes: 2 points, often: 3 points, and almost always: 4 points. Minimum and maximum scores of the inventory are 17 points and 68 points, respectively. Higher scores indicate that severity of fatigue increases. A score of 25 or more from the inventory indicates the presence of depression. At this cut-off point, the sensitivity and specificity of the inventory are 97% and 86%. The Cronbach's alpha value of the inventory is 0.893. The inventory has four subscales; low mood subscale: 7 items (7-28 points), inhibition of movement and thought subscale: 4 items (4-16 points), change in cognition subscale: 4 items (4-16 points), low self-evaluation subscale: 2 items (2-8 points). Higher scores mean that the situation reflected by the subscale worsens.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Assoc. Prof., Principal Investigator — Istanbul University
Locations (1):
- Nurten Ozen, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang YY, Zhang WW, Feng L, Gao D, Liu C, Zhong L, Ren JW, Wu YZ, Huang L, Fu LL, He YN. Development and Preliminary Validation of a Depression Assessment Tool for Maintenance Hemodialysis Patients. Ther Apher Dial. 2019 Feb;23(1):49-58. doi: 10.1111/1744-9987.12749. Epub 2018 Sep 21. PMID 30239119
- [Result] Palmer S, Vecchio M, Craig JC, Tonelli M, Johnson DW, Nicolucci A, Pellegrini F, Saglimbene V, Logroscino G, Fishbane S, Strippoli GF. Prevalence of depression in chronic kidney disease: systematic review and meta-analysis of observational studies. Kidney Int. 2013 Jul;84(1):179-91. doi: 10.1038/ki.2013.77. Epub 2013 Mar 13. PMID 23486521